CLINICAL TRIAL: NCT06657521
Title: Influence of the Osteoimplant Vitamin Complex on the Stability of Dental Implants. Randomized Double-blind Clinical Trial.
Brief Title: Osteoimplant and Dental Implants Stability
Acronym: OIMP
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Francisco Javier Manzano-Moreno, PhD, Doctor in Dental Surgery, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4054/CEIH/2024
Record Dates: First submitted 2024-10-23; First posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Primary Stability of the Implants; Pain
Keywords: Dental implant; vitamin c; vitamin D; stability; pain; inflamation
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OSTEOIMPLANT GROUP (Experimental): patients prescribed to take Osteoimplant Complex© on the following schedule: 2 tablets per day starting 5 days before implant placement and 1 tablet per day of Osteimplant© for 2 months after implant placement.
  Interventions: Dietary Supplement: osteoimplant
- Placebo Group (Placebo Comparator): 30 patients who were prescribed placebo with the following regimen: 2 tablets per day starting 5 days before implant placement and 1 tablet per day for 2 months after implant placement.
  Interventions: Dietary Supplement: Placebo Oral Tablet

INTERVENTIONS:
Dietary Supplement: osteoimplant — Osteoimplant Complex© on the following schedule: 2 tablets per day starting 5 days before implant placement and 1 tablet per day of Osteimplant© for 2 months after implant placement.
  Arms: OSTEOIMPLANT GROUP
Dietary Supplement: Placebo Oral Tablet — 2 tablets per day starting 5 days before implant placement and 1 tablet per day for 2 months after implant placement.
  Arms: Placebo Group

SUMMARY:
Based on the scientific evidence, the relevance of this subject, we consider this study to be justified, the general or specific objective of which is as follows:

'To evaluate the effect of the administration of Osteoimplant© and Osteoimplant Complex© as a food supplement in obtaining implant stability and in the healing of dental implant surgery'.

As secondary objectives, we will also evaluate the effect of Osteoimplant© and Osteoimplant Complex© on pain, postoperative inflammation and soft tissue healing.

The sample will consist of 60 patients. The sample will be randomly divided into 2 groups using a randomisation table generated by a statistical programme. For blinding, neither the patient nor the operator shall be aware of the group to which each patient belongs. To ensure blinding, medication will be delivered in sealed, opaque envelopes. Patients shall be assigned to one of the following groups:

* Group I: 30 patients prescribed to take Osteoimplant Complex© on the following schedule: 2 tablets per day starting 5 days before implant placement and 1 tablet per day of Osteimplant© for 2 months after implant placement.
* Group II: 30 patients who were prescribed placebo with the following regimen: 2 tablets per day starting 5 days before implant placement and 1 tablet per day for 2 months after implant placement.

DETAILED DESCRIPTION:
Based on the scientific evidence, the relevance of this subject, we consider this study to be justified, the general or specific objective of which is as follows:

'To evaluate the effect of the administration of Osteoimplant© and Osteoimplant Complex© as a food supplement in obtaining implant stability and in the healing of dental implant surgery'.

As secondary objectives, we will also evaluate the effect of Osteoimplant© and Osteoimplant Complex© on pain, postoperative inflammation and soft tissue healing.

The sample will consist of 60 patients. The sample will be randomly divided into 2 groups using a randomisation table generated by a statistical programme. For blinding, neither the patient nor the operator shall be aware of the group to which each patient belongs. To ensure blinding, medication will be delivered in sealed, opaque envelopes. Patients shall be assigned to one of the following groups:

* Group I: 30 patients prescribed to take Osteoimplant Complex© on the following schedule: 2 tablets per day starting 5 days before implant placement and 1 tablet per day of Osteimplant© for 2 months after implant placement.
* Group II: 30 patients who were prescribed placebo with the following regimen: 2 tablets per day starting 5 days before implant placement and 1 tablet per day for 2 months after implant placement.

3.1. Study design Our study is a double-blind randomised clinical trial (RCT) to evaluate the stability of the implants in the different phases of treatment: at the time of insertion (primary stability), at 8 and 12 weeks (secondary stability). Postoperative pain and swelling will also be studied.

Composition of nutritional supplements.

* The preoperative nutritional supplement corresponds to Osteoimplant Complex® and is composed of: vitamin C 48.5 mg, coenzyme Q10 41.3 mg, Zinc 35 mg, beta-carotene 10% 25 mg, bioflavonoids citrus 60% 20.83 mg, vitamin E and magnesium 15 mg.
* The post-operative nutritional supplement corresponds to Osteoimplant®, and is composed of: Ovocet ®, collagen 350 mg, calcium 300 mg, vitamin D3 100IU/mg, magnesium 8 mg.

Patients Conceptual or target population Patients with partial or total single tooth edentulism requiring rehabilitation with intraosseous implants.

Study or accessible population The patients who will form part of our study will be those who attend the Master's Degree in Oral Surgery and Implantology of the Faculty of Dentistry of the University of Granada requesting dental implants for their rehabilitation.

All patients will undergo a clinical history and subsequent clinical examination. The clinical history will consist of an anamnesis, where the patient's personal details will be collected (name, age, sex, profession, address and telephone number), as well as family history, illnesses suffered, previous surgical interventions, drug allergies and current treatment. Subsequently, an intraoral and extraoral examination will be carried out, consisting of inspection and palpation of the bucco-facial territory.

To complement our examination and make a correct diagnosis, all patients will undergo a radiological study as a step prior to surgery, which will always consist of an orthopantomography, the usual projection for this type of intervention, with which a correct diagnosis can be made. In addition, we will complete the study with a CBCT in order to assess three-dimensionally the relationship with anatomical structures and the availability of bone.

Once the diagnosis has been correctly made, the patient will be informed, both orally and in writing, of the possible complications that may arise in this type of surgery. The following inclusion and exclusion criteria will be applied to the target population for participation in the study:

Inclusion criteria:

* Patients presenting with unitary or partial edentulism.
* Age: Between 18-75 years.
* Anaesthetic risk ASA I-II.
* Patients who do not abuse alcohol, drugs or chronic smoking (>10 cigarettes/day).
* Patients with adequate periodontal status (≤10% plaque index and bleeding index).
* Absence of drug allergies that could compromise our study.
* Absence of allergy to any of the components of Osteoimplant© and Osteimplant Complex©.
* Signed informed consent.

Exclusion criteria:

* Age not between 18-75 years old.
* Pregnant or breastfeeding women.
* Chronic smokers (>10 cigarettes/day).
* Patients with decompensated metabolic disease.
* Poor periodontal status (≥10% plaque index and bleeding index).
* Patients allergic to any of the components of Osteoimplant© and Osteimplant Complex©.
* Patients undergoing treatment with drugs that could affect the bone regeneration process, such as chemotherapy drugs, bisphosphonates, corticosteroids or immunosuppressants.
* Patients with metabolic bone diseases or who have undergone radiotherapy in the last five years.
* Patients with hypercalcaemia or a tendency to hypercalcification, taking vitamin D or calcium supplements.
* Patients with a history of renal colic.
* Patients who are not going to undergo nephrotic colic. 1. Surgical Protocol First of all, the patient rinses with 0.12% chlorhexidine. After 1 minute, the area to be implanted is anaesthetised using a truncal block or infiltrative technique with 4% articaine together with epinephrine. A transcrestal or paracrestal incision is made, depending on the case, and the mucoperiosteal flap is detached. Once detached, the position of the implant will be determined thanks to the in situ visualisation of the bone thickness and the previous CBCT study of each patient. Subsequently, the drilling sequence is determined by the company itself. Once the implant bed has been created, we will proceed to insert the implant with a torque of at least 30-45N. At this point, the first stability measurement will be taken, then the cover screw will be placed and the flap and suture will be repositioned. The patient will be reviewed and given a series of postoperative guidelines in physical format, which it is essential to follow for a correct result of our surgery.

All implants will be placed following the same surgical protocol and in strict compliance with the implant manufacturer's instructions regarding the drilling protocol associated with the patient's bone quality.

Once the implants are placed, stability measurements shall be taken with the Osstell ISQ and the stability levels of the implants shall be evaluated at different stages of treatment by performing the following measurements:

1. First measurement: after implant placement surgery. We will evaluate the primary stability.
2. Second measurement: at 8 weeks to determine the evolution of osseointegration throughout the healing process of our implants.
3. Third measurement: at 12 weeks to assess the evolution of osseointegration again before subjecting the implant to occlusal loads.

Prior to implant placement, each patient will be assigned to a study group, where, depending on their assignment, they will receive either placebo or the drug in question:

Preoperative phase:

* Group I: prescribed to take Osteoimplant Complex ® 2 every 24 hours, 5 days prior to surgery.
* Group II: prescribed to take placebo 2 every 24 hours, 5 days prior to surgery.

Post-operative phase:

* Group I: prescribed to take Osteoimplant® 1 every 24 hours, for 8 weeks after surgery.
* Group II: prescribed placebo 1 every 24 hours for 8 weeks after surgery. In both groups, an antibiotic treatment of amoxicillin 500 mg, 1 every 8 hours for 5 days is administered. In case of penicillin allergy, the drug of choice will be clindamycin 300 mg 1 every 8 hours for 5 days; as well as an analgesic and anti-inflammatory treatment: ibuprofen 400 mg 1 every 8 hours for 2 days, from the third day on demand. As rescue medication paracetamol 1 g.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with unitary or partial edentulism.

  * Age: Between 18-75 years.
  * Anaesthetic risk ASA I-II.
  * Patients who do not abuse alcohol, drugs or chronic smoking (>10 cigarettes/day).
  * Patients with adequate periodontal status (≤10% plaque index and bleeding index).
  * Absence of drug allergies that could compromise our study.
  * Absence of allergy to any of the components of Osteoimplant© and Osteimplant Complex©.
  * Signed informed consent.

Exclusion Criteria:

* Age not between 18-75 years old.
* Pregnant or breastfeeding women.
* Chronic smokers (>10 cigarettes/day).
* Patients with decompensated metabolic disease.
* Poor periodontal status (≥10% plaque index and bleeding index).
* Patients allergic to any of the components of Osteoimplant© and Osteimplant Complex©.
* Patients undergoing treatment with drugs that could affect the bone regeneration process, such as chemotherapy drugs, bisphosphonates, corticosteroids or immunosuppressants.
* Patients with metabolic bone diseases or who have undergone radiotherapy in the last five years.
* Patients with hypercalcaemia or a tendency to hypercalcification, taking vitamin D or calcium supplements.
* Patients with a history of renal colic.
* Patients who are not going to undergo nephrotic colic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
IMPLANT STABILITY | From implant placement until 12 weeks
  All implants will be placed following the same surgical protocol and in strict compliance with the implant manufacturer's instructions regarding the drilling protocol associated with the patient's bone quality.
  Once the implants are placed, stability measurements shall be taken with the Osstell ISQ and the stability levels of the implants shall be evaluated at different stages of treatment by performing the following measurements:
  1. First measurement: after implant placement surgery. We will evaluate the primary stability.
  2. Second measurement: at 8 weeks to determine the evolution of osseointegration throughout the healing process of our implants.
  3. Third measurement: at 12 weeks to assess the evolution of osseointegration again before subjecting the implant to occlusal loads.
  Prior to implant placement, each patient will be assigned to a study group, where, depending on their assignment, they will receive either placebo or the drug in question:

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Chen MH, Lyons KM, Tawse-Smith A, Ma S. Clinical Significance of the Use of Resonance Frequency Analysis in Assessing Implant Stability: A Systematic Review. Int J Prosthodont. 2019 Jan/Feb;32(1):51-58. doi: 10.11607/ijp.6048. PMID 30677112
- [Result] Werny JG, Sagheb K, Diaz L, Kammerer PW, Al-Nawas B, Schiegnitz E. Does vitamin D have an effect on osseointegration of dental implants? A systematic review. Int J Implant Dent. 2022 Apr 11;8(1):16. doi: 10.1186/s40729-022-00414-6. PMID 35403929
- [Result] Dermience M, Lognay G, Mathieu F, Goyens P. Effects of thirty elements on bone metabolism. J Trace Elem Med Biol. 2015 Oct;32:86-106. doi: 10.1016/j.jtemb.2015.06.005. Epub 2015 Jun 26. PMID 26302917
- [Result] Choi HK, Kim GJ, Yoo HS, Song DH, Chung KH, Lee KJ, Koo YT, An JH. Vitamin C Activates Osteoblastogenesis and Inhibits Osteoclastogenesis via Wnt/beta-Catenin/ATF4 Signaling Pathways. Nutrients. 2019 Feb 27;11(3):506. doi: 10.3390/nu11030506. PMID 30818817
- [Result] Kim JH, Lim YJ, Kim B, Lee J. How Do Parameters of Implant Primary Stability Correspond with CT-Evaluated Bone Quality in the Posterior Maxilla? A Correlation Analysis. Materials (Basel). 2021 Jan 7;14(2):270. doi: 10.3390/ma14020270. PMID 33430383